CLINICAL TRIAL: NCT03576885
Title: Treatment of Delayed Pulmonary Transition in Extremely Preterm Infants & Bronchopulmonary Dysplasia
Brief Title: Inhaled Nitric Oxide for Pulmonary Hypertension and Bronchopulmonary Dysplasia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: based on DSMB recommendation at interim analysis
Sponsor: AdventHealth (Other)
Collaborators: Mallinckrodt (Industry); Thrasher Research Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1170748
Record Dates: First submitted 2018-06-22; First posted 2018-07-03 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Hypertension; Bronchopulmonary Dysplasia
MeSH Terms: conditions — Hypertension, Pulmonary; Bronchopulmonary Dysplasia

STUDY DESIGN:
Intervention Model Description: Masked randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment group - active (Active Comparator): inhaled nitric oxide treatment will start at 20 ppm and continue for 2 weeks or until resolution of pulmonary hypertension, whichever comes first.
  Interventions: Drug: inhaled nitric oxide
- Treatment group - placebo (Placebo Comparator): Placebo treatment will start at 20 ppm and continue for 2 weeks or until resolution of pulmonary hypertension, whichever comes first.
  Interventions: Drug: Placebo
- Control group (No Intervention): Enrolled infants with no evidence of pulmonary hypertension will serve as the control group for incidence of death or bronchopulmonary hypertension

INTERVENTIONS:
Drug: inhaled nitric oxide — inhaled nitric oxide will be administered starting at 20 ppm. Treatment will continue for 14 days or until resolution of pulmonary hypertension
  Other Names: iNO
  Arms: Treatment group - active
Drug: Placebo — placebo will be administered starting at 20 ppm. Treatment will continue for 14 days or until resolution of pulmonary hypertension
  Arms: Treatment group - placebo

SUMMARY:
Inhaled nitric oxide (iNO) is an effective treatment for pulmonary hypertension (PH) in term and near-term infants. Preterm infants are at risk for early PH that is associated with high risk for bronchopulmonary dysplasia or death. In multiple clinical trials, iNO treatment was not effective for BPD prevention. However, infants were not screened for PH and iNO treatment was not targeted for PH. iNO treatment for PH in preterm infants is controversial due to lack of evidence. The study team hypothesizes that early diagnosis of PH (72-96 hours of life) and iNO treatment will decrease the incidence of death and bronchopulmonary dysplasia and improve oxygenation in extremely preterm infants.

1. To determine if iNO treatment of extremely preterm infants with early pulmonary hypertension as established with echocardiographic evidence at 72-96 hours of age will decrease incidence of death or BPD.
2. To determine if iNO treatment of extremely preterm infants with early PH will decrease the pulmonary artery pressure and improve oxygenation within 72 hours of intervention.

DETAILED DESCRIPTION:
This is a single center, blinded, randomized control clinical trial to evaluate the effects of inhaled nitric oxide on the outcome of survival and incidence of bronchopulmonary dysplasia. This trial has a planned enrollment of 138 infants with 68 infants with delayed pulmonary transition assigned to either the treatment or placebo group. There is no enrollment restriction based on gender, ethnicity, or race. Enrollment is expected to take 36 months with an additional 12 months for data analysis.Infants with early pulmonary hypertension will be randomized to the treatment or placebo group. Treatment will continue until resolution of pulmonary hypertension or through Day 14, whichever comes first. Serial echocardiograms will be performed every 48 hours +/-12 hours until Day 14. Oxygen saturation levels will be averaged every 24 hour period following enrollment. This study will provide evidence for the beneficial effects of early diagnosis and treatment of pulmonary hypertension in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

Step 1:

* Birth between 23 weeks and 0 days and 29 weeks and 6 days.
* Positive pressure ventilation at 72-96 hours of age

Step 2:

* Early pulmonary hypertension

Exclusion Criteria:

Step 1:

* Death prior to 12 hours of age or first echocardiogram
* Chromosomal anomalies
* Major congenital anomalies
* Myocardial dysfunction
* Complex cardiac defect
* Dependent on right to left shunting of blood

Step 2:

* Excessive pulmonary blood flow (left to right shunt across PDA)
* Pulmonary blood flow obstruction secondary to pulmonary vein stenosis
* Mitral valve stenosis
* Cor triata
* Aortic valve atresia

Ages: 23 Weeks to 29 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2023-10-09 (Actual); Study Completion 2023-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hussnain Mirza, MD, Principal Investigator — AdventHealth
Locations (1):
- AdventHealth, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Laughon MM, Langer JC, Bose CL, Smith PB, Ambalavanan N, Kennedy KA, Stoll BJ, Buchter S, Laptook AR, Ehrenkranz RA, Cotten CM, Wilson-Costello DE, Shankaran S, Van Meurs KP, Davis AS, Gantz MG, Finer NN, Yoder BA, Faix RG, Carlo WA, Schibler KR, Newman NS, Rich W, Das A, Higgins RD, Walsh MC; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Prediction of bronchopulmonary dysplasia by postnatal age in extremely premature infants. Am J Respir Crit Care Med. 2011 Jun 15;183(12):1715-22. doi: 10.1164/rccm.201101-0055OC. Epub 2011 Mar 4. PMID 21471086
- [Background] Ballard RA, Keller RL, Black DM, Ballard PL, Merrill JD, Eichenwald EC, Truog WE, Mammel MC, Steinhorn RH, Rogers EE, Ryan RM, Durand DJ, Asselin JM, Bendel CM, Bendel-Stenzel EM, Courtney SE, Dhanireddy R, Hudak ML, Koch FR, Mayock DE, McKay VJ, O'Shea TM, Porta NF, Wadhawan R, Palermo L; TOLSURF Study Group. Randomized Trial of Late Surfactant Treatment in Ventilated Preterm Infants Receiving Inhaled Nitric Oxide. J Pediatr. 2016 Jan;168:23-29.e4. doi: 10.1016/j.jpeds.2015.09.031. Epub 2015 Oct 21. PMID 26500107
- [Background] Khemani E, McElhinney DB, Rhein L, Andrade O, Lacro RV, Thomas KC, Mullen MP. Pulmonary artery hypertension in formerly premature infants with bronchopulmonary dysplasia: clinical features and outcomes in the surfactant era. Pediatrics. 2007 Dec;120(6):1260-9. doi: 10.1542/peds.2007-0971. PMID 18055675
- [Background] West JB, Mathieu-Costello O. Stress failure of pulmonary capillaries as a limiting factor for maximal exercise. Eur J Appl Physiol Occup Physiol. 1995;70(2):99-108. doi: 10.1007/BF00361536. PMID 7768245
- [Background] Mirza H, Ziegler J, Ford S, Padbury J, Tucker R, Laptook A. Pulmonary hypertension in preterm infants: prevalence and association with bronchopulmonary dysplasia. J Pediatr. 2014 Nov;165(5):909-14.e1. doi: 10.1016/j.jpeds.2014.07.040. Epub 2014 Sep 1. PMID 25189821
- [Background] Bhat R, Salas AA, Foster C, Carlo WA, Ambalavanan N. Prospective analysis of pulmonary hypertension in extremely low birth weight infants. Pediatrics. 2012 Mar;129(3):e682-9. doi: 10.1542/peds.2011-1827. Epub 2012 Feb 6. PMID 22311993
- [Background] Mourani PM, Sontag MK, Younoszai A, Miller JI, Kinsella JP, Baker CD, Poindexter BB, Ingram DA, Abman SH. Early pulmonary vascular disease in preterm infants at risk for bronchopulmonary dysplasia. Am J Respir Crit Care Med. 2015 Jan 1;191(1):87-95. doi: 10.1164/rccm.201409-1594OC. PMID 25389562
- [Background] Ambalavanan N, Mourani P. Pulmonary hypertension in bronchopulmonary dysplasia. Birth Defects Res A Clin Mol Teratol. 2014 Mar;100(3):240-6. doi: 10.1002/bdra.23241. Epub 2014 Mar 10. PMID 24616323
- [Background] Finer NN, Evans N. Inhaled nitric oxide for the preterm infant: evidence versus practice. Pediatrics. 2015 Apr;135(4):754-6. doi: 10.1542/peds.2015-0144. Epub 2015 Mar 9. No abstract available. PMID 25755239
- [Background] Kinsella JP, Steinhorn RH, Krishnan US, Feinstein JA, Adatia I, Austin ED, Rosenzweig EB, Everett AD, Fineman JR, Hanna BD, Hopper RK, Humpl T, Ivy DD, Keller RL, Mullen MP, Raj JU, Wessel DL, Abman SH. Recommendations for the Use of Inhaled Nitric Oxide Therapy in Premature Newborns with Severe Pulmonary Hypertension. J Pediatr. 2016 Mar;170:312-4. doi: 10.1016/j.jpeds.2015.11.050. Epub 2015 Dec 15. No abstract available. PMID 26703869
- [Background] Abman SH, Kinsella JP, Schaffer MS, Wilkening RB. Inhaled nitric oxide in the management of a premature newborn with severe respiratory distress and pulmonary hypertension. Pediatrics. 1993 Oct;92(4):606-9. No abstract available. PMID 8414836
- [Background] Ambalavanan N, Aschner JL. Management of hypoxemic respiratory failure and pulmonary hypertension in preterm infants. J Perinatol. 2016 Jun;36 Suppl 2:S20-7. doi: 10.1038/jp.2016.45. PMID 27225961
- [Background] Askie LM, Ballard RA, Cutter GR, Dani C, Elbourne D, Field D, Hascoet JM, Hibbs AM, Kinsella JP, Mercier JC, Rich W, Schreiber MD, Wongsiridej PS, Subhedar NV, Van Meurs KP, Voysey M, Barrington K, Ehrenkranz RA, Finer NN; Meta-analysis of Preterm Patients on Inhaled Nitric Oxide Collaboration. Inhaled nitric oxide in preterm infants: an individual-patient data meta-analysis of randomized trials. Pediatrics. 2011 Oct;128(4):729-39. doi: 10.1542/peds.2010-2725. Epub 2011 Sep 19. PMID 21930540
- [Background] Truog WE, Ballard PL, Norberg M, Golombek S, Savani RC, Merrill JD, Parton LA, Cnaan A, Luan X, Ballard RA; Nitric Oxide (to Prevent) Chronic Lung Disease Study Investigators. Inflammatory markers and mediators in tracheal fluid of premature infants treated with inhaled nitric oxide. Pediatrics. 2007 Apr;119(4):670-8. doi: 10.1542/peds.2006-2683. PMID 17403837
- [Background] Posencheg MA, Gow AJ, Truog WE, Ballard RA, Cnaan A, Golombek SG, Ballard PL; NO CLD Investigators. Inhaled nitric oxide in premature infants: effect on tracheal aspirate and plasma nitric oxide metabolites. J Perinatol. 2010 Apr;30(4):275-80. doi: 10.1038/jp.2009.155. Epub 2009 Oct 8. PMID 19812581
- [Background] Mourani PM, Abman SH. Pulmonary Hypertension and Vascular Abnormalities in Bronchopulmonary Dysplasia. Clin Perinatol. 2015 Dec;42(4):839-55. doi: 10.1016/j.clp.2015.08.010. Epub 2015 Sep 26. PMID 26593082
- [Background] Kumar P; Committee on Fetus and Newborn; American Academy of Pediatrics. Use of inhaled nitric oxide in preterm infants. Pediatrics. 2014 Jan;133(1):164-70. doi: 10.1542/peds.2013-3444. Epub 2013 Dec 30. PMID 24379225
- [Background] Cole FS, Alleyne C, Barks JD, Boyle RJ, Carroll JL, Dokken D, Edwards WH, Georgieff M, Gregory K, Johnston MV, Kramer M, Mitchell C, Neu J, Pursley DM, Robinson W, Rowitch DH. NIH consensus development conference: Inhaled nitric oxide therapy for premature infants. NIH Consens State Sci Statements. 2010 Oct 29;27(5):1-34. PMID 21042341
- [Background] Abman SH, Hansmann G, Archer SL, Ivy DD, Adatia I, Chung WK, Hanna BD, Rosenzweig EB, Raj JU, Cornfield D, Stenmark KR, Steinhorn R, Thebaud B, Fineman JR, Kuehne T, Feinstein JA, Friedberg MK, Earing M, Barst RJ, Keller RL, Kinsella JP, Mullen M, Deterding R, Kulik T, Mallory G, Humpl T, Wessel DL; American Heart Association Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation; Council on Clinical Cardiology; Council on Cardiovascular Disease in the Young; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular Surgery and Anesthesia; and the American Thoracic Society. Pediatric Pulmonary Hypertension: Guidelines From the American Heart Association and American Thoracic Society. Circulation. 2015 Nov 24;132(21):2037-99. doi: 10.1161/CIR.0000000000000329. Epub 2015 Nov 3. PMID 26534956
- [Background] Seth SA, Soraisham AS, Harabor A. Risk factors and outcomes of early pulmonary hypertension in preterm infants. J Matern Fetal Neonatal Med. 2018 Dec;31(23):3147-3152. doi: 10.1080/14767058.2017.1365129. Epub 2017 Aug 21. PMID 28783986
- [Background] Jiang Q, Gao X, Liu C, Chen D, Lin X, Xia S, Zhuang D, Yang C, Zhu W, Liu L, Chen C, Sun B. Early inhaled nitric oxide in preterm infants <34 weeks with evolving bronchopulmonary dysplasia. J Perinatol. 2016 Oct;36(10):883-9. doi: 10.1038/jp.2016.112. Epub 2016 Jul 21. PMID 27442155
- [Background] Mercier JC, Hummler H, Durrmeyer X, Sanchez-Luna M, Carnielli V, Field D, Greenough A, Van Overmeire B, Jonsson B, Hallman M, Baldassarre J; EUNO Study Group. Inhaled nitric oxide for prevention of bronchopulmonary dysplasia in premature babies (EUNO): a randomised controlled trial. Lancet. 2010 Jul 31;376(9738):346-54. doi: 10.1016/S0140-6736(10)60664-2. Epub 2010 Jul 23. PMID 20655106
- [Background] Kinsella JP, Cutter GR, Steinhorn RH, Nelin LD, Walsh WF, Finer NN, Abman SH. Noninvasive inhaled nitric oxide does not prevent bronchopulmonary dysplasia in premature newborns. J Pediatr. 2014 Dec;165(6):1104-1108.e1. doi: 10.1016/j.jpeds.2014.06.018. Epub 2014 Jul 22. PMID 25063725
- [Background] Evans N. Towards rational use of inhaled Nitric Oxide in preterm babies. Acta Paediatr. 2016 Feb;105(2):121-2. doi: 10.1111/apa.13273. No abstract available. PMID 26751417
- [Background] Arul N, Konduri GG. Inhaled nitric oxide for preterm neonates. Clin Perinatol. 2009 Mar;36(1):43-61. doi: 10.1016/j.clp.2008.09.002. PMID 19161864
- [Background] Giesinger RE, More K, Odame J, Jain A, Jankov RP, McNamara PJ. Controversies in the identification and management of acute pulmonary hypertension in preterm neonates. Pediatr Res. 2017 Dec;82(6):901-914. doi: 10.1038/pr.2017.200. Epub 2017 Oct 4. PMID 28820870
- [Background] Mirza H, Garcia JA, Crawford E, Pepe J, Zussman M, Wadhawan R, Oh W. Natural History of Postnatal Cardiopulmonary Adaptation in Infants Born Extremely Preterm and Risk for Death or Bronchopulmonary Dysplasia. J Pediatr. 2018 Jul;198:187-193.e1. doi: 10.1016/j.jpeds.2018.02.034. Epub 2018 Apr 3. PMID 29625730
- [Background] Bilan N, Dastranji A, Ghalehgolab Behbahani A. Comparison of the spo2/fio2 ratio and the pao2/fio2 ratio in patients with acute lung injury or acute respiratory distress syndrome. J Cardiovasc Thorac Res. 2015;7(1):28-31. doi: 10.15171/jcvtr.2014.06. Epub 2015 Mar 29. PMID 25859313
- [Background] Pandharipande PP, Shintani AK, Hagerman HE, St Jacques PJ, Rice TW, Sanders NW, Ware LB, Bernard GR, Ely EW. Derivation and validation of Spo2/Fio2 ratio to impute for Pao2/Fio2 ratio in the respiratory component of the Sequential Organ Failure Assessment score. Crit Care Med. 2009 Apr;37(4):1317-21. doi: 10.1097/CCM.0b013e31819cefa9. PMID 19242333
- [Background] Peliowski A; Canadian Paediatric Society, Fetus and Newborn Committee. Inhaled nitric oxide use in newborns. Paediatr Child Health. 2012 Feb;17(2):95-100. doi: 10.1093/pch/17.2.95. PMID 23372402

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group - Active | Treatment Group - Placebo | Control Group
Started | 16 | 16 | 0
Completed | 16 | 16 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group - Active | Treatment Group - Placebo | Control Group | Total
Number analyzed (Participants) | 16 | 16 | 0 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 16 | 0 | 32
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: days] | 3 (1) | 3 (1) |  | 3 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 0 | 10
  Male | 11 | 11 | 0 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 7 | 0 | 14
  White | 7 | 8 | 0 | 15
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 16 | 0 | 32

OUTCOME MEASURES:

1. Primary Outcome: Death
Description: Incidence of death
Time Frame: 36 weeks post menstrual age
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group - Active | Treatment Group - Placebo
Number analyzed (Participants) | 16 | 16
Participants | 1 | 1

2. Primary Outcome: Bronchopulmonary (BPD) Dysplasia (Yes/no)
Description: Incidence of bronchopulmonary dysplasia as determined by need for positive pressure ventilation or supplemental oxygen after room air challenge test
Time Frame: 36 weeks post menstrual age
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group - Active | Treatment Group - Placebo
Number analyzed (Participants) | 16 | 16
Participants | 10 | 9

3. Secondary Outcome: Pulmonary Hypertension
Description: Pulmonary arterial pressure will be evaluated every 24-48 hours after enrollment.
Time Frame: Duration of treatment or up to Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group - Active | Treatment Group - Placebo
Number analyzed (Participants) | 16 | 16
Participants | 11 | 15

ADVERSE EVENTS:
Time Frame: Until 36 weeks post-menstrual age
Arm/Group | Treatment Group - Active | Treatment Group - Placebo
All-Cause Mortality (participants affected / at risk) | 1/16 | 1/16
Serious Adverse Events (participants affected / at risk) | 2/16 | 5/16
Other Adverse Events (participants affected / at risk) | 14/16 | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group - Active (N=16) | Treatment Group - Placebo (N=16)
IVH (Nervous system disorders) | 2 (2) | 2 (2) — Intraventricular Hemorrhage
NEC (Gastrointestinal disorders) | 0 (0) | 3 (3) — Necrotizing Enterocolitis
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group - Active (N=16) | Treatment Group - Placebo (N=16)
MetHb% >2 (Blood and lymphatic system disorders) | 3 (3) | 5 (5) — Methemoglobinemia
Culture positive sepsis (Infections and infestations) | 5 (5) | 9 (9) — Culture proven sepsis treated with antibiotics
PDA requiring treatment (Cardiac disorders) | 3 (3) | 4 (4) — Patent ductus arteriosus requiring medical or surgical treatment
Left Ventricular Dysfunction (Cardiac disorders) | 1 (1) | 1 (1) — Left ventricular dysfunction or EF less than 40%
Hyperbilirubinemia (Hepatobiliary disorders) | 7 (7) | 7 (7) — Neonatal Jaundice treated by Phototherapy
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) — Platelets less than 100,000

LIMITATIONS AND CAVEATS:
Majority of preterm infants with hypoxic respiratory failure or severe pulmonary hypertension were excluded due to the clinical treatment with inhaled nitric oxide prior to our study echocardiogram

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/85/NCT03576885/Prot_SAP_000.pdf